CLINICAL TRIAL: NCT00728377
Title: An Exercise Intervention to Prevent Recurrent GDM
Brief Title: An Exercise Intervention to Prevent Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Lisa Chasan-Taber, Professor, University of Massachusetts, Amherst
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DK74876; R01DK074876 (NIH); 1R01DK074876-01A1 (NIH); NCT01141582 (obsolete NCT alias)
Record Dates: First submitted 2008-08-02; First posted 2008-08-05 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Gestational Diabetes
Keywords: gestational diabetes; physical activity; behavior change; glucose tolerance; pregnancy
MeSH Terms: conditions — Diabetes, Gestational; Motor Activity | interventions — Exercise; Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heath & Wellness (Active Comparator)
  Interventions: Behavioral: Heath & Wellness
- Exercise (Experimental)
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Physical activity — Individually Tailored (IT) Exercise Intervention This intervention is designed to increase the amount of physical activity incorporated into the daily lifestyle of pregnant women, primarily through increased walking, with the ultimate goal of achieving the American College of Obstetricians and Gynecologists (ACOG) exercise goals for pregnant women. These goals are the same as the Surgeon General's Guidelines for physical activity for nonpregnant individuals (30 minutes or more or moderate activity on most days of the week).The intervention includes: 1) individually tailored print-based materials (i.e., individually-tailored reports and stage-matched manuals), 2) self-monitoring materials, and 3) goal setting.
  Arms: Exercise
Behavioral: Heath & Wellness — The comparison intervention consists of a series of informational booklets published by the American College of Obstetricians and Gynecologists on general issues related to health and wellness during pregnancy. These include alcohol and drug use during pregnancy, easing back pain, as well as the Pregnancy Fitness brochure on the safety of exercise during pregnancy. These booklets are selected to represent high-quality, standard, low-cost, self-help material currently available to the public.
  Arms: Heath & Wellness

SUMMARY:
Women diagnosed with gestational diabetes mellitus (GDM) are at substantially increased risk of developing type 2 diabetes and obesity, currently at epidemic rates in the United States. GDM, therefore, identifies a population of women at high risk of developing type 2 diabetes and thus provides an excellent opportunity to intervene years before the development of this disorder. It is well recognized that acute as well as chronic physical activity reduce fasting plasma glucose as well as improve glucose tolerance in type 2 diabetes. Recent studies have suggested that women with higher levels of physical activity have reduced risk of GDM. Therefore, we will test the hypothesis that an exercise intervention is an effective tool for preventing GDM among women with a history of GDM.

DETAILED DESCRIPTION:
The primary goals of the application are to investigate the effects of a motivationally-tailored, individually targeted 12-wk physical activity intervention on 1) risk of GDM in women at high risk of the condition, 2) serum biomarkers associated with insulin resistance, 3) and the adoption and maintenance of exercise during pregnancy. Secondary goals are to investigate the impact of the intervention on gestational weight gain and selected birth outcomes. The overall goal of the intervention is to encourage pregnant women to achieve the American College of Obstetricians and Gynecologists (ACOG) Guidelines for physical activity during pregnancy (30 minutes or more of moderate- intensity activity on most days of the week) through increasing walking and developing a more active lifestyle. The intervention draws from the theory of Stages of Motivational Readiness for Change and Social Cognitive Theory constructs for physical activity behavior and will take into account the specific social, cultural, economic, and physical environmental challenges faced by women of diverse socioeconomic and ethnic backgrounds. The application is innovative in being the first, to our knowledge, to test a physical activity intervention designed to prevent GDM among high risk women. The intervention protocol can readily be translated into clinical practice in underserved and minority populations.

ELIGIBILITY:
Inclusion Criteria:

* history of gestational diabetes or overweight (>25 kg/m2) with family history of type 2 diabetes
* sedentary

Exclusion Criteria:

* history of diagnosis of diabetes, hypertension, heart disease or chronic renal disease
* current medications which adversely influence glucose tolerance
* not planning to continue the pregnancy to term
* >16 weeks gestation
* contraindications to participating in moderate physical activity
* inability to read English at a 6th grade level
* self-reported participation in >30 min of moderate or vigorous-intensity exercise on >3 days/wk
* prior participation in the study
* non-singleton pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 488 (Actual)
Dates: Start 2007-07; Primary Completion 2011-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Gestational diabetes diagnosis assessed through glucose tolerance test. | 28 weeks gestational age

SECONDARY OUTCOMES:
Maternal weight gain | 40 weeks gestational age
Glucose | 28 weeks gestational age
Insulin | 28 weeks gestational age
Adiponectin | 28 weeks gestational age
Resistin | 28 weeks gestational age
TNF-alpha | 28 weeks gestational age
CRP | 28 weeks gestational age
Birth weight | 40 weeks gestational age
Apgar score | 40 weeks gestational age
Adoption and maintenance of exercise during pregnancy | 40 weeks gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Chasan-Taber, Principal Investigator — University of Massachusetts, Amherst
Locations (1):
- Batstate Medical Center, Springfield, Massachusetts, United States

REFERENCES:
- [Background] Hawkins M, Chasan-Taber L, Marcus B, Stanek E, Braun B, Ciccolo J, Markenson G. Impact of an exercise intervention on physical activity during pregnancy: the behaviors affecting baby and you study. Am J Public Health. 2014 Oct;104(10):e74-81. doi: 10.2105/AJPH.2014.302072. Epub 2014 Aug 14. PMID 25122031
- [Derived] Hawkins M, Braun B, Marcus BH, Stanek E 3rd, Markenson G, Chasan-Taber L. The impact of an exercise intervention on C - reactive protein during pregnancy: a randomized controlled trial. BMC Pregnancy Childbirth. 2015 Jun 24;15:139. doi: 10.1186/s12884-015-0576-2. PMID 26104503
- [Derived] Nobles C, Marcus BH, Stanek EJ 3rd, Braun B, Whitcomb BW, Solomon CG, Manson JE, Markenson G, Chasan-Taber L. Effect of an exercise intervention on gestational diabetes mellitus: a randomized controlled trial. Obstet Gynecol. 2015 May;125(5):1195-1204. doi: 10.1097/AOG.0000000000000738. PMID 25932848
- [Derived] Chasan-Taber L, Silveira M, Marcus BH, Braun B, Stanek E, Markenson G. Feasibility and efficacy of a physical activity intervention among pregnant women: the behaviors affecting baby and you (B.A.B.Y.) study. J Phys Act Health. 2011 Sep;8 Suppl 2(0 2):S228-38. PMID 21918237